CLINICAL TRIAL: NCT02779309
Title: An Algorithm for Predicting Death Among Older Adults in the Home Care Setting: Study Protocol for the Risk Evaluation for Support: Predicting Elder Life in the Community Tool (RESPECT)
Brief Title: Risk Evaluation for Support: Predicting Elder Life in the Community Tool (RESPECT)
Acronym: RESPECT
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Institute for Clinical Evaluative Sciences (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: CIHR FRN - 142876; Trim no. P0901 074 (Other: Institute for Clinical Evaluative Sciences)
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Death
Keywords: Frail Older Adults; Mortality; Home Care; Survival Analysis; Clinical Prediction Rule
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Development Cohort: 437,000 home care recipients who received services from January 1, 2007 to December 31, 2012.
  Interventions: Procedure: Home Care/RAI-HC Assessment
- Validation Cohort: 122,000 home care recipients who received services from January 1, 2013 to December 31, 2013.
  Interventions: Procedure: Home Care/RAI-HC Assessment

INTERVENTIONS:
Procedure: Home Care/RAI-HC Assessment — Home care recipients who have received a comprehensive health assessment using the Resident Assessment Instrument for Home Care (RAI-HC).

SUMMARY:
To develop a mortality risk prediction model that can be applied to the wide spectrum of risks that are seen in the home care setting.

DETAILED DESCRIPTION:
ABSTRACT

Introduction: Older adults living in the community often have multiple, chronic conditions and functional impairments. A challenge for healthcare providers working in the community is the lack of a predictive tool that can be applied to the broad spectrum of mortality risks observed and may be used to inform care planning.

Objective: To develop a mortality risk prediction model for older adults in the home care setting. The final algorithm will be implemented as a web-based calculator that can be used by older adults needing care, as well as their informal and formal caregivers.

Design: Open cohort study using the Resident Assessment Instrument for Home Care (RAI-HC) data in Ontario, Canada, from January 1, 2007, to December 31, 2013.

Participants: The derivation cohort will consist of approximately 437 000 home care recipients from January 1, 2007, to December 31, 2012. A split sample validation cohort will include approximately 122 000 recipients from January 1 to December 31, 2013.

Main outcome measures: Predicted survival from the time of an RAI-HC assessment. All deaths (N ≈ 245 000) will be ascertained through linkage to the provincial vital statistics records.

Statistical analysis: Proportional hazards regression will be estimated after assessment of assumptions. Predictors will include sociodemographic characteristics, social support, health conditions, functional status, cognition, symptoms of decline, and prior healthcare use. Model performance will be evaluated for 6- and 12-month predicted risks, including measures of calibration (e.g., calibration plots) and discrimination (e.g., c-statistics). The final algorithm will be generated by combining development and validation data.

ELIGIBILITY:
Inclusion Criteria:

* Have received a structured RAI-HC assessment
* Between 50 and 105 years of age

Exclusion Criteria:

* Not eligible for Ontario's universal health insurance program (OHIP)
* Did not receive a structured RAI-HC assessment

Ages: 50 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older adults receiving home care in Ontario, Canada, who have received a structured Resident Assessment Instrument for Home Care (RAI-HC) assessment between January 1, 2007 and December 31, 2013.
Sampling Method: Non-Probability Sample
Enrollment: 486000 (Actual)
Dates: Start 2007-01; Primary Completion 2013-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
6-month Mortality | 6 months
  Mortality status at 6 months after receiving a structured Resident Assessment Instrument for Home Care (RAI-HC) Assessment.

SECONDARY OUTCOMES:
12-month Mortality | 12 months
  Mortality status at 12 months after receiving a structured Resident Assessment Instrument for Home Care (RAI-HC) Assessment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu AT, Manuel DG, Taljaard M, Chalifoux M, Bennett C, Costa AP, Bronskill S, Kobewka D, Tanuseputro P. Algorithm for predicting death among older adults in the home care setting: study protocol for the Risk Evaluation for Support: Predictions for Elder-life in the Community Tool (RESPECT). BMJ Open. 2016 Dec 1;6(12):e013666. doi: 10.1136/bmjopen-2016-013666. PMID 27909039